CLINICAL TRIAL: NCT01779830
Title: A Randomized, Double-Blind, Placebo-Controlled, Dose-Ranging, Crossover Study of Single Doses of LY2624803 in a 5-hour Phase Advance Model of Transient Insomnia in Healthy Subjects
Brief Title: A Study of LY2624803 in Participants With Transient Insomnia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: 12057; I2K-MC-ZZAA (Other: Eli Lilly and Company)
Record Dates: First submitted 2013-01-25; First posted 2013-01-30 (Estimated); Last update posted 2013-01-30 (Estimated); Status verified 2013-01

CONDITIONS: Transient Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Zolpidem

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- 0.3 mg LY2624803 (Experimental): Single dose of 0.3 mg LY2624803 administered orally in up to 2 of 4 treatment periods.
  Interventions: Drug: LY2624803 - Capsules
- 3.0 mg LY2624803 (Experimental): Single dose of 3.0 mg LY2624803 administered orally in up to 2 of 4 treatment periods.
  Interventions: Drug: LY2624803 - Capsules
- 6.0 mg LY2624803 (Experimental): Single dose of 6.0 mg LY2624803 administered orally in up to 2 of 4 treatment periods.
  Interventions: Drug: LY2624803 - Capsules
- 10 mg Zolpidem (Active Comparator): Single dose of 10 mg zolpidem administered orally in up to 1 of 4 treatment periods.
  Interventions: Drug: Zolpidem - Tablets
- Placebo (Placebo Comparator): Single dose of placebo administered orally in up to 1 of 4 treatment periods.
  Interventions: Drug: Placebo - Capsules; Drug: Placebo - Tablets

INTERVENTIONS:
Drug: LY2624803 - Capsules — Administered orally as capsules.
  Other Names: Hypnion
  Arms: 0.3 mg LY2624803; 3.0 mg LY2624803; 6.0 mg LY2624803
Drug: Zolpidem - Tablets — Administered orally as tablets.
  Arms: 10 mg Zolpidem
Drug: Placebo - Capsules — Administered orally as capsules.
  Arms: Placebo
Drug: Placebo - Tablets — Administered orally as tablets.
  Arms: Placebo

SUMMARY:
The aim of this study is to learn how different doses of LY2624803 affect sleep in healthy people. The study has four treatment periods. Participants will receive a single dose of LY2624803, another sleeping pill, or placebo in each treatment period. The study will last approximately 1 month for each participant.

ELIGIBILITY:
Inclusion Criteria:

* Overtly healthy males or females
* Women of child-bearing potential, who test negative for pregnancy at the time of enrollment based on a urine pregnancy test and agree to use a reliable method of birth control during the study and for one month following the last dose of study drug
* Between the Body Mass Index (BMI) of 19 and 30 kilogram per meter square (kg/m^2), inclusive
* Normal bedtime hours, with routine time spent in bed between 6.5 hours and 9 hours each night
* Participants whose daily caffeine intake permits maintenance of normal bed time hours
* Non response to placebo defined as a Wake After Sleep Onset (WASO) of greater than or equal to 45 minutes, on a 5-hour phase-advanced polysomnography (PSG) screening night after bedtime single-blind placebo administration
* Males must agree to use effective barrier contraception during the course of the trial and 3 months later
* Participants over 65 years of age, on a stable dose of one medication for lowering cholesterol, triglycerides and/or one medication for lowering blood pressure and/or substitutive hormonal therapy in post menopausal women are allowed provided those treatments have no central effect
* Clinical laboratory test results within normal reference range judged to be not clinically significant
* Normal sitting blood pressure and pulse rate as determined
* Venous access sufficient to allow blood sampling
* Are reliable and willing to make themselves available for the duration of the study
* Have given written informed consent approved by Lilly and the ethical review board governing the site

Exclusion Criteria:

* Shift workers (those who shifted work within 7 days of any PSG night) or any person who has crossed (or will have crossed) more than one time zone by aircraft within 3 days prior to entry
* Rhinoconjunctivitis, urticaria or chronic pain severe enough to interfere with sleep
* Nocturia that would interfere with sleep assessment
* Participants with allergic conjunctivitis or urticaria
* Regular napping (greater than (≥) 2 daytime naps/week by history)
* Symptoms consistent with a sleep disorder or history of same
* Sleep disorders detected during the screening night
* Evidence of significant active neuropsychiatric disease and in particular evidence of significant medical or psychiatric illness within the past 12 months that could contribute to insomnia
* Irregular or altered sleep/wake schedule
* Known history of fainting or low blood pressure. History of cranial trauma and loss of consciousness will be discussed prior to including any such participant
* Within 3 months of the initial dose of study drug, have received treatment with a drug that has not received regulatory approval for any indication
* Participants with postural hypotension at screening
* Participants with a history of postural hypotension, loss of consciousness, explained or unexplained syncope or seizure episodes or a family history of seizures. History of a single febrile convulsion is acceptable
* Known allergies to LY2624803, Zolpidem or related compounds
* Persons who have previously completed or withdrawn from this study or any other study investigating LY2624803
* An abnormality in the 12-lead electrocardiogram (ECG) that increases the risks associated with participating in the study
* History or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, neurocardiogenic or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; of constituting a risk when taking the study medication; or of interfering with the interpretation of data
* Any other condition with in the opinion of the investigator would preclude participation the study
* Regular use of known drugs of abuse and/or positive findings on urinary drug screening
* Evidence of Human Immunodeficiency Virus (HIV) and/or positive human HIV antibodies
* Evidence of hepatitis C and/or positive hepatitis C antibody
* Evidence of hepatitis B and/or positive hepatitis B surface antigen
* Women with a positive pregnancy test
* Women who are lactating
* Use of prescription, over the counter or herbal medications that cannot safely be discontinued within 28 days prior to enrollment
* Blood donation of more than 500 milliliter (mL) within the last month
* History of smoking within the previous 6 months of screening
* Participants who have an average weekly alcohol intake that exceeds 28 units per week (males) and 21 units per week (females), or participants unwilling to stop alcohol consumption for the duration of the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2008-05; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Change in Wake After Sleep Onset (WASO) With LY2624803 Compared to Placebo | Baseline up to Day 60

SECONDARY OUTCOMES:
Latency to Persistent Sleep (LPS) with LY2624803 Compared to Placebo | Baseline up to Day 60
Total Sleep Time (TST) with LY2624803 Compared to Placebo | Baseline up to Day 60

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rouffach, France